CLINICAL TRIAL: NCT06931470
Title: A Pilot Feasibility and Acceptability Study of Remote ExerciSe Training mOdalities
Brief Title: A Pilot Feasibility and Acceptability Study of Remote ExerciSe Training mOdalities (PRESTO)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-01067
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- In-Person Supervised Aerobic Exercise Intervention (IPSAEI) (Active Comparator): Participants engage in supervised exercise sessions at a facility, where trainers use centralized telemetry to monitor heart rates and provide immediate feedback and adjustments to exercise intensity.
  Interventions: Behavioral: In-person supervised exercise sessions; Device: Centralized telemetry
- Remote Synchronous Aerobic Exercise Intervention (RSAEI) (Experimental): Participants join live-streamed exercise sessions led by a virtual trainer. Real-time heart rate monitoring via an app allows the trainer to provide immediate feedback and adjust exercise intensity as needed.
  Interventions: Behavioral: Virtual classes (live-streamed sessions); Device: Map My Fitness mobile application
- Asynchronous Remote Aerobic Exercise Intervention (RASAEI) (Experimental): Participants exercise independently while monitoring their heart rate in real time using the Map My Fitness app. They adjust their intensity based on personal targets and receive periodic feedback from a trainer during scheduled check-ins.
  Interventions: Behavioral: Self-directed aerobic exercise; Device: Map My Fitness mobile application
- Remote MyZone Aerobic Exercise Intervention (RMZAEI) (Experimental): Participants use the Myzone heart rate monitor and app to receive real-time feedback on their exercise intensity. The Myzone platform provides automated guidance on intensity adjustments, goal setting, and motivational support through features like challenges and social connectivity.
  Interventions: Device: Myzone mobile application; Device: Myzone heart rate monitor

INTERVENTIONS:
Behavioral: In-person supervised exercise sessions — Gold-standard, facility-based sessions (3 sessions/week) with an onsite trainer guidance with an exercise Intensity of 40-80% heart rate reserve (HRR) or Rate of Perceived Exertion (RPE) 12-16.
  Arms: In-Person Supervised Aerobic Exercise Intervention (IPSAEI)
Behavioral: Virtual classes (live-streamed sessions) — Live-streamed exercise classes (3 sessions/week) with a trainer providing real-time feedback.
  Arms: Remote Synchronous Aerobic Exercise Intervention (RSAEI)
Behavioral: Self-directed aerobic exercise — Participants exercise independently and follow a weekly progression plan (3-5 sessions/week (depending on the specific progression)).
  Arms: Asynchronous Remote Aerobic Exercise Intervention (RASAEI)
Device: Myzone mobile application — Training using the Myzone platform, with participants wearing the Myzone heart rate monitor and using the Myzone app to receive real-time feedback and guidance during exercise sessions (3 days per week). Myzone integrates with its proprietary wearable devices to monitor heart rate and other activity metrics, providing real-time data to users via the app.
  Arms: Remote MyZone Aerobic Exercise Intervention (RMZAEI)
Device: Map My Fitness mobile application — Participants will wear a Bluetooth-compatible heart rate monitor (e.g., apple watch/fitbit) that syncs with MapMyFitness. MapMyFitness automatically records workout sessions (duration, distance, heart rate, calories burned, and elevation gain where applicable).
  Arms: Asynchronous Remote Aerobic Exercise Intervention (RASAEI); Remote Synchronous Aerobic Exercise Intervention (RSAEI)
Device: Centralized telemetry — Centralized telemetry monitors heart rates and provides immediate feedback for trainers to adjust exercise intensity.
  Arms: In-Person Supervised Aerobic Exercise Intervention (IPSAEI)
Device: Myzone heart rate monitor — Wearable device (chest strap or armband) that monitors heart rate.
  Arms: Remote MyZone Aerobic Exercise Intervention (RMZAEI)

SUMMARY:
This study will investigate the acceptability and efficacy of 12 weeks of: Smart-device app-based (MyZone) Asynchronous Virtual, Synchronous Virtual, and in-person aerobic training in individuals at risk for Cardiovascular Disease (CVD) who do are not meeting American Heart Association (AHA) guidelines for physical activity. The study aims to 1) Assess the effect of several approaches to remote aerobic training on measures of physical activity, cardiovascular fitness and CVD risk, and 2) Quantitatively and qualitatively evaluate exercise training program fidelity, implementation, effectiveness, and remaining barriers to acceptance.

Participants will be asked to undergo Cardiopulmonary Exercise Testing (CPET) before and after 12-weeks of training via one of the 4 modalities (random assignment) listed above. They will respond to questions regarding acceptability of the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. >45 years
2. At risk for CVD (participants must have one or more of the following risk factors: hypertension, hyperlipidemia, Type 2 Diabetes Mellitus, smoking, obesity, family history of premature CVD)
3. Not meeting AHA physical activity guidelines for at least 3 months prior to screening

   * Hypertension:

     * Systolic BP ≥140 mm Hg and/or diastolic BP ≥90 mm Hg and/or
     * Use of anti-hypertensive medication
   * Hyper / dyslipidemia

     * LDL cholesterol levels ≥160 mg/dL and/or
     * HDL cholesterol <50mg/dL for women, <40mg/dL for women, in addition to fasting triglycerides >150mg/dL
   * Diabetes Mellitus:

     * Hemoglobin A1c levels ≥6.5%, fasting glucose levels ≥126 mg/dL, or 2-hour glucose levels ≥200 mg/dL after an oral glucose tolerance test and/or
     * Use of any diabetes medication
   * Smoking:

     o Current regular tobacco use.
   * Obesity:

     o BMI ≥30 kg/m².
   * Family History of Premature Cardiovascular Disease:

     * Having a first-degree relative (parent, sibling) who developed CVD before age 55 for biological males or age 65 for biological females.

Exclusion Criteria:

1. Established diagnosis of atherosclerotic CVD
2. Presence of any serious medical conditions that would not allow safe participation in exercise according to the American College of Sports Medicine (ACSM) and the AHA (56-58)
3. Pregnant or anticipating pregnancy
4. Plan to be away for >2 weeks during the intervention period
5. Presence of any biopsychosocial factors that the principal investigator deems as having significant potential to interfere with effective study participation

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Average minutes of moderate to vigorous physical activity per week | Up to 13 weeks
  Outcome is measured via wearable technology (smart device).

SECONDARY OUTCOMES:
Change in peak oxygen consumption (VO2peak) | Baseline, Week 13
  Peak oxygen consumption (VO2peak) is measured as the highest VO2 recorded during the course of a Cardiopulmonary Exercise Testing (CPET).
Change in blood pressure | Baseline, Week 13
Change in Body mass index (BMI) | Baseline, Week 13
  BMI (kg/m2) will be calculated using measured body weight and height
Change in body fat percentage | Baseline, Week 13
  Body fat percentage will be assessed via multi-frequency bioelectrical impedance analysis (BIA) with 8 tactile electrodes.
Change in fasting glucose levels | Baseline, Week 13
Change in 36-Item Short Form Survey Instrument (SF-36) | Baseline, Week 13
  SF-36 captures mental health, general health perception, emotional, and social role functioning. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. Higher scores indicate a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P. Heffron, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: [Alec Sinatro, MD; alec.sinatro@nyulangone.org]. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to [Alec Sinatro, MD; alec.sinatro@nyulangone.org]. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.